CLINICAL TRIAL: NCT01517672
Title: Neurobiology of Severe Psychological Trauma in Women
Brief Title: Imaging Outcomes of Cognitive Behavioral Therapy (CBT) for Battered Women With Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Murray B. Stein, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: STEIN VA MERIT
Record Dates: First submitted 2012-01-16; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; domestic violence; intimate partner violence; functional MRI; neuroimaging
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive Trauma Therapy for Battered Women (CTT-BW) — 10 individual sessions of this form of cognitive therapy, with a trained therapist.

SUMMARY:
Identifying neural mechanisms of posttraumatic stress disorder (PTSD) treatment could help elucidate reasons for variable treatment response and identify novel treatment targets. Exposure-based therapies have been associated with decreased amygdala and increased cingulate cortex response during emotional processing. The current study examined whether cognitive therapy for PTSD in women reduces activation in insula and amygdala and enhances activation in prefrontal regions during emotional anticipation and pre-treatment prefrontal activation predicts treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Intimate partner violence (IPV) trauma defined as physical and/or sexual abuse committed by a romantic partner, occurring within five years of, but having ended at least one month prior to, enrollment in the study.
* Seeking treatment for posttraumatic stress disorder (PTSD) symptoms and meeting full or partial Diagnostic and Statistical Manual, 4th edition (DSM-IV) criteria for PTSD prior to treatment, verified through the Clinician-Administered PTSD Scale (CAPS).

Exclusion Criteria:

* Substance abuse in the past year
* History of >2 years of alcohol abuse
* Use of psychotropic medications within 4 weeks prior to the study, bipolar disorder or schizophrenia, irremovable ferromagnetic bodily material, pregnancy, or claustrophobia.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS) | After 10 sessions of cognitive behavioral therapy (CBT) (10-14 weeks)
  The CAPS is a widely used measure of PTSD severity. Intent was to administer 10 sessions of CBT over a period of 10-14 weeks. Primary outcome was CAPS at the end of CBT administration.

SECONDARY OUTCOMES:
CAPS 3 months post-treatment | 3 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Murray B Stein, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States